CLINICAL TRIAL: NCT00408213
Title: A Randomized, Double-Blind Study to Evaluate the Safety of Continued Treatment With CellCept in Patients With Well-Controlled Myasthenia Gravis Receiving a Stable Dose of Prednisone
Brief Title: A Continuation Study to Assess the Effect of CellCept in Patients With Myasthenia Gravis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Aspreva Pharmaceuticals (Industry)
Responsible Party: Clinical Trials, Study Director, Hoffmann-La Roche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WX18411; NCT00231088 (obsolete NCT alias)
Record Dates: First submitted 2006-12-05; First posted 2006-12-06 (Estimated); Last update posted 2008-05-23 (Estimated); Status verified 2008-05

CONDITIONS: Myasthenia Gravis Generalised
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: mycophenolate mofetil [CellCept]
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept] — 1g po bid
  Arms: 1
Drug: Placebo — po bid
  Arms: 2

SUMMARY:
This 2 arm study will provide optional continuation of double-blind treatment with CellCept or placebo, in patients with myasthenia gravis who have achieved good symptom control in study WX17798. Patients who have completed 36 weeks of treatment in study WX17798, with stable prednisone dosing for the last 4 weeks, can continue on blinded treatment with CellCept (1g bid) or placebo until the database for WX17798 is locked and unblinded. The anticipated time on study treatment is 3-12 months, and the target sample size is 100-500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* subjects who have completed 36 weeks of treatment in study WX17798, and who have demonstrated good symptom control with a stable prednisone dose for the final 4 weeks of that study.

Exclusion Criteria:

* regularly scheduled plasma exchange or intravenous immunoglobulin treatment;
* medical condition, adverse event or intolerance of double-blind treatment which would preclude continuation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2004-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, vital signs. | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (3):
  - Sun City, Arizona
  - Sacramento, California
  - Upland, Pennsylvania
- France (2):
  - Bordeaux
  - Nice
- Germany (2):
  - München
  - Regensburg
- Italy (2):
  - Milan
  - Roma
- Belgrade, Serbia and Montenegro
- Ukraine (3):
  - Kharkiv
  - Kiev
  - Zaporizhzhya
- United Kingdom (3):
  - Liverpool
  - Oxford
  - Salford